CLINICAL TRIAL: NCT01266941
Title: An Open-label, Non-randomized, Pharmacokinetic and Safety Study of Repeat Doses of Fluticasone Furoate and GW642444M Combination in Healthy Subjects and in Subjects With Mild, Moderate or Severe Hepatic Impairment
Brief Title: A Study to Assess the Effects of Fluticasone Furoate and GW642444M Combination in Healthy Subjects and in Subjects With Mild, Moderate or Severe Hepatic Impairment.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 111789
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Asthma
Keywords: pharmacokinetics; hepatic impairment; heart rate; serum potassium; serum cortisol; GW642444M; Fluticasone furoate (GW685698)
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mild Hepatic Impairment (Experimental): Mild and moderate hepatic patients will be recruited first, approximately 9 subjects should complete each of these treatment arms.
  Interventions: Drug: Inhaled FF 200mcg/GW642444M 25mcg
- Moderate Hepatic Impairment (Experimental): Mild and moderate hepatic patients will be recruited first, approximately 9 subjects should complete each of these treatment arms.
  Interventions: Drug: Inhaled FF 200mcg/GW642444M 25mcg
- Matched healthy volunteers (Experimental): Once a moderate subject has been recruited, a healthy control subject should be recruited (matched to the moderate subject on gender, ethnicity, body mass index +/-15%, age +/-5 years). In total there will be 9 matched healthy volunteers 1 for each subject with moderate hepatic impairment.
  Interventions: Drug: Inhaled FF 200mcg/GW642444M 25mcg
- Severe Hepatic Impairment (Experimental): Severe subjects will not be enrolled into the study until 9 moderate subjects and their matched control subjects have completed the study and the safety and PK data have been reviewed.
  Interventions: Drug: Inhaled FF 200mcg/GW642444M 25mcg

INTERVENTIONS:
Drug: Inhaled FF 200mcg/GW642444M 25mcg — All subjects are scheduled to receive FF 200mcg/GW642444M 25mcg once daily for 7 days. The dose for subjects with severe hepatic impairment may be adjusted to FF 100mcg/GW642444M 12.5mcg after review of the PK and safety data from the moderate and healthy matched control subjects.

SUMMARY:
In relation to their severity, hepatic diseases can significantly modify drug absorption and disposition and consequently can interfere with drug efficacy and/or produce toxicity. The purpose of this study will be to aid in deciding whether a dose adjustment is required in subjects with hepatic impairment and in estimating any such adjustments.

DETAILED DESCRIPTION:
In relation to their severity, hepatic diseases can significantly modify drug absorption and disposition and consequently can interfere with drug efficacy and/or produce toxicity. Pathological modifications of liver structure or functionality might result in complex modifications of various factors including liver blood flow, hypoalbuminaemia, indirectly affect renal function and reduce the hepatic drug metabolizing capability including the microsomal oxidase system [Howden, 1989].

Although FF/GW642444M is delivered directly to the site of action, i.e. the lungs, a large portion of the administered dose is swallowed. For both FF and GW642444 any drug absorbed from the GI tract undergoes first pass metabolism via CYP3A4. In addition, drug absorbed into the systemic circulation is metabolised in the liver and removed by biliary clearance. Hence, there is a possibility that when used by patients with impaired liver function the pharmacokinetics of inhaled FF and/or GW642444 may be changed due to reduced first pass metabolism and/or reduced clearance. The results of this study will aid in deciding whether a dose adjustment is justified and in estimating any such adjustments in patients with impaired hepatic function.

This is an open-label, non-randomized study which will assess the pharmacokinetics and safety of inhaled FF 200mcg/GW642444M 25mcg in subjects with hepatic impairment following 7 days once daily dosing. Subjects with mild, moderate and severe hepatic impairment (as defined by a Child-Pugh score of 5-15) will be recruited along with healthy control subjects matched to the moderate subjects (matched on gender, ethnicity, body mass index +/-15%, age +/-5 years).

Approximately thirty-six subjects will be recruited: 9 subjects for each severity and 9 matched healthy subjects. All subjects are scheduled to receive FF 200mcg/GW642444M 25mcg once daily for 7 days. The dose for subjects with severe hepatic impairment may be adjusted to FF 100mcg/GW642444M 12.5mcg after review of the PK and safety data from the moderate and healthy matched control subjects. The results of this study will aid in deciding whether a dose adjustment is required in subjects with hepatic impairment and in estimating any such adjustments.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

* Male or female between 18 and 70 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of:

  * Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) (healthy subjects only) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
  * Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until completion of the follow-up visit.
* BMI within the range 19 - 33 kg/m^2.
* Able to satisfactorily use the dry powder inhalation inhaler.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Single QTcF < 450 msec; or QTcF < 480 msec in subjects with Bundle Branch Block.
* Able to satisfactorily use the dry powder inhaler.

Healthy subjects:

* AST, ALT, alkaline phosphatase and bilirubin ≤1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures or outcome.

Hepatically Impaired Subjects:

- Hepatically impaired.

To be classified as hepatically impaired, subjects must have:

Known medical history of liver disease with or without a known history of alcohol abuse; and A Child-Pugh score of 5-15 to cover all severities (Mild = 5-6 points; Moderate = 7-9 points; Severe = 10-15 points). The components that contribute to the CP score should be directly related to the underlying hepatic disease and not to non-hepatic disease.

- Subjects with no significant abnormality, apart from impaired hepatic function and related symptoms, or clinical examination. A subject with a clinical abnormality may be included only if the Investigator considers that the abnormality will not introduce additional risk factors and will not interfere with the study procedures. Hepatically impaired subjects with other laboratory parameters outside the reference ranges will only be included if, in the opinion of the Investigator, the result is not clinically important and introduces no additional risk factors.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Suffered a lower respiratory tract infection in the 4 weeks before the screening visit.
* Taken oral corticosteroids less than 8 weeks before the screening visit.
* Taken inhaled, intranasal or topical steroids less than 4 weeks before the screening visit.
* Have a known sensitivity to corticosteroids and/or long acting beta agonists.
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.
* The subject has been treated for or diagnosed with depression within six months of screening or has a history of significant psychiatric illness.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Subjects who have asthma or a history of asthma.
* History of severe milk protein allergy.
* Subjects with a smoking history of >10 cigarettes per day or regular use of tobacco- or nicotine-containing products, within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Healthy subjects

* If, in the opinion of the examining physician, an unstable cardiovascular, renal, hepatic, pulmonary, endocrine, metabolic, neurological, haematological or gastrointestinal condition is present or any other medical condition which the investigator considers sufficiently serious to interfere with the conduct, completion, or results of this trial or constitutes an unacceptable risk to the subject.
* Subjects with any predisposing condition that might interfere with the absorption, distribution, metabolism or excretion of drugs or any previous gastrointestinal (GI) surgery (except appendectomy or cholecystectomy more than three months prior to the study) condition which the investigator considers sufficiently significant to interfere with the conduct, completion, or results of this trial or constitutes an unacceptable risk to the subject.
* Haemoglobin values <12.9g/dL for males and <11.4g/dL for females.
* A past history or current symptoms of significant hepatic or renal disease, pancreatitis or acute cholecystitis which the investigator considers sufficiently significant to interfere with the conduct, completion, or results of this trial or constitutes an unacceptable risk to the subject.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as:

  • An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inhibitor) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety. In particular subjects taking steroids or medications that significantly inhibit P450 CYP3A4 (e.g. ketoconazole) must not be included in this study.

Hepatically Impaired Subjects

* If in the opinion of the examining physician, an unstable cardiovascular, renal, pulmonary, endocrine, metabolic, neurological, haematological or gastrointestinal condition is present or any other significant medical condition which the investigator considers sufficiently serious to interfere with the conduct, completion, or results of this trial or constitutes an unacceptable risk to the subject.
* Severe ascities (Child-Pugh ascites score of 3) upon clinical exam, including physical exam and abdominal ultrasound at screening. Subjects identified to have moderate ascities by ultrasound examination may be included at the discretion of the Investigator with prior agreement from the sponsor.
* History of oesophageal bleeding within the last 6 months before dosing.
* Significant hepatic encephalopathy, degree of CNS impairment or other signs of hepatic function deterioration which the investigator considers sufficiently serious to interfere with the informed consent, conduct, completion, or results of this trial or constitutes an unacceptable risk to the subject.
* Patients at risk of requiring a transfusion during the study period, or has haemoglobin < 9 g/dL, or has underlying coronary artery disease (or other clinical condition) in which a reduction in haemoglobin associated with FF/GW642444M administration might be expected to cause clinical deterioration.
* Evidence of current significant infection (e.g. spontaneous bacterial peritonitis, pneumonia etc.).
* Subjects who develop symptoms such as infections or haemorrhage between screening and dosing must not be included in the study.
* Fluctuating or rapidly deteriorating hepatic function (such as, but not limited to, rapidly increasing ascites, rapidly deteriorating mental status, deteriorating hepatic function based on prothrombin time [PT], albumin, total bilirubin). Assessment of the stability of the subject's hepatic function will be at the discretion of the Principal Investigator.
* Subjects with significant renal insufficiency as defined by estimated creatinine clearance of <50 ml/min, using the Cockcroft and Gault equation.
* Subjects with a diagnosis of primary biliary disease such as cholestasis or sclerosing cholangitis.
* Subjects who need to take any concomitant medication, either prescribed or over-the-counter, which may in the opinion of the Investigator, interfere in any way with the study procedure or be a safety concern (see Section 9 for the list of permitted concurrent medications). In particular subjects taking medications that significantly inhibit P450 CYP3A4 (e.g. ketoconazole) must not be included in this study.
* Subjects who, within the past six months, have had a history of significant drug abuse or alcohol abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-10-18 (Actual); Primary Completion 2011-07-15 (Actual); Study Completion 2011-07-15 (Actual)

PRIMARY OUTCOMES:
Fluticasone furoate and GW642444 pharmacokinetics (AUC(0-t), AUC (0-8), Cmax, tmax) on Day 1 and 7 and AUC(0-24) and t½ on Day 7. | 1 Month

SECONDARY OUTCOMES:
Serum cortisol weighted mean over 24 hours on Days -1 and 7. | 1 Month
Maximum heart rate over time period 0-4 hours on Day 7. | 1 Month
Minimum serum potassium concentration over time period 0-4 hours on Day 7. | 1 Month
General safety and tolerability endpoints: adverse events, blood pressure, heart rate, 12-lead ECG, clinical laboratory safety tests. | 1 Month

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Czechia (2):
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Prague
- GSK Investigational Site, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Allen A, Davis A, Hardes K, Tombs L, Kempsford R. Influence of renal and hepatic impairment on the pharmacokinetic and pharmacodynamic properties and tolerability of fluticasone furoate and vilanterol in combination. Clin Ther. 2012 Dec;34(12):2316-32. doi: 10.1016/j.clinthera.2012.11.001. Epub 2012 Nov 30. PMID 23200625
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 111789 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/111789?search=study&study_ids=111789#rs
- Available data/document: Annotated Case Report Form: 111789 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111789 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111789 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111789 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111789 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111789 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111789 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register